CLINICAL TRIAL: NCT04414254
Title: Bioequivalence of Cefprozil for Suspension and Granule Formulation in Healthy Chinese Volunteers: Two Single-Dose Crossover Studies
Brief Title: Bioequivalence of Cefprozil Granule in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-YK1-036-001
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Cefprozil; Suspensions

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, single-dose, two-period, two-group, crossover study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conference-Cefprozil for Suspension® (Experimental): "Cefprozil for Suspension®" (125mg/5ml, 50ml/bottle, batch no. F701087, manufactured by Lupin Pharmaceuticals, Inc.)
  Interventions: Drug: Cefprozil 125mg/5ml Susp; Cefprozil granule (125mg)
- test-cefprozil granule (Experimental): cefprozil granule (125mg, batch no. 8G001F07, manufactured by Qilu Pharmaceutical Co., Ltd)
  Interventions: Drug: Cefprozil 125mg/5ml Susp; Cefprozil granule (125mg)

INTERVENTIONS:
Drug: Cefprozil 125mg/5ml Susp; Cefprozil granule (125mg) — Subjects were allocated to one of two groups randomly and equally with a 3-day washout interval between the two periods."Cefprozil for Suspension®" (125mg/5mL, 50mL/bottle, batch no. F701087, manufactured by Lupin Pharmaceuticals, Inc.) and cefprozil granule (125mg, batch no. 8G001F07, manufactured by Qilu Pharmaceutical Co., Ltd) were used in this study.

SUMMARY:
An open-label, randomized, single-dose, two-period, two-group, crossover study was conducted in 60 healthy Chinese volunteers under fasted or fed conditions (30 volunteers for each condition) to assess the bioequivalence between two formulations of cefprozil.

DETAILED DESCRIPTION:
Cefprozil, an oral second-generation semi-synthetic cephalosporin, possesses a broad spectrum of antimicrobial activity. A granule formulation has been developed to improve medication adherence of the patients. This study was conducted to assess the bioequivalence of the granule formulation to dry suspension in healthy Chinese volunteers and estimate the pharmacokinetics profiles of cefprozil. An open-label, randomized, single-dose, two-period, two-group, crossover study was conducted in 60 healthy Chinese volunteers under fasted or fed conditions (30 volunteers for each condition) to assess the bioequivalence between two formulations of cefprozil. Blood samples were collected at specified time intervals, and the plasma concentrations of cis- and trans-cefprozil were determined by a validated liquid chromatography- mass spectrum/ mass spectrum method. Pharmacokinetic and bioavailability parameters were estimated via non-compartmental methods. Adverse events were also recorded. If the 90% confidence intervals of the ratios of geometrical mean of test and reference formulations for Cmax, AUC0-t and AUC0-infer are all within the predefined bioequivalence criteria range of 80%-125% for cis-, trans-and total cefprozil, the two formulations can be considered bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged between 18 and 55 years old (including the critical value).
* The body mass index is in the range of 19-28 kg/m2 (including the critical value). The weight of male is not less than 50 kg, and that of female is not less than 45 kg (including the critical value).
* Subjects who had not any medical history of cardiovascular, digestive, respiratory, nervous, haemal diseases or hepatic/renal impairment.The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: physical examination, 12-lead ECG, vital sign measurements, and laboratory safety tests .
* The subjects have no family planning within 6 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.
* The subjects could complete the study accorrding to the protocol.

Exclusion Criteria:

* any history of hypersensitivity, needlesickness or idiosyncratic reactions to any food or drug, especially for penicillins or cephalosporins;
* hepatitis (including hepatitis B and C), positive screening results for AIDS or syphilis;
* any history of acute or chronic illness that might affect drug absorption, and/or metabolism;
* positive results for urine drug screening;
* any history of drug abuse in the past 5 years or drug use 3 months prior to screening;
* any history of alcohol abuse in the recent 2 years or moderate drinkers (drink more 2 units per day or 14 units per week);
* smoking more than 5 cigarettes per day during the 3 months prior to screening;
* blood donation, massive blood loss (>400mL) or enrolled in other clinical trials 3 months prior to screening;
* any use of other prescription drugs (including contraceptive) 14 days prior to medication for this study;
* any use of prescription or over-the-counter drugs, functional vitamin, herbal/ alcohol products, grapefruit-containing or caffeine/xanthine-rich foodand beverages 48 h prior to medication for this study;
* the outcome of breath alcohol test > 0mg /mL;
* dysphagia or having special dietary requirements;
* occurring acute disease in the screening period or before the medication;
* lactating or pregnant women;
* investigator-determined ineligibility.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
the ratios of geometrical mean | 71 Days
  The two preparations were considered bioequivalent if the 90% CIs of the ratios of the primary pharmacokinetics parameters were within the predefined acceptance range of 80%-125%.

SECONDARY OUTCOMES:
the occurrence rate of adverse events | 71 Days
  Adverse events were recorded to evaluate the safety of the studied drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by Qilu Pharmaceutical Co., Ltd. and the research center. The research center can not publish any academic papers without the consent of the sponsor.

REFERENCES:
- [Derived] Lin PP, Wang CJ, Liu YP, Li T, Gao XM, Ma YP, Shi P, Li X, Wang LX, Cao Y. Pharmacokinetics and Bioequivalence of Cefprozil for Suspension and Granule Formulation in Healthy Chinese Volunteers: Two Single-Dose Crossover Studies. Adv Ther. 2021 Feb;38(2):1130-1142. doi: 10.1007/s12325-020-01593-7. Epub 2020 Dec 19. PMID 33340343